CLINICAL TRIAL: NCT00000920
Title: A Phase I Trial of the Safety and Pharmacokinetics of Fortovase (Saquinavir-SGC) Co-Administered With Low Dose (Ritonavir) RTV, ZDV and 3TC in HIV Seropositive Pregnant Women During Gestation and Postpartum, and in Their Infant's Post-Maternal Dosing
Brief Title: Fortovase (Saquinavir) Given With Low-Dose Ritonavir, Zidovudine, and Lamivudine to HIV-Positive Pregnant Women During and After Pregnancy and to Their Newborns
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: ACTG 386; 11345 (Registry Identifier: DAIDS ES); PACTG 386
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Drug Therapy, Combination; Zidovudine; Pregnancy Complications; Ritonavir; Lamivudine; Saquinavir; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Pregnancy Complications | interventions — Ritonavir; Saquinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Ritonavir
Drug: Saquinavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if it is safe to give saquinavir-SGC (SQV) combined with low-dose ritonavir (RTV) plus zidovudine (ZDV) and lamivudine (3TC) to HIV-positive pregnant women and to see if it is safe to give 3TC and ZDV to their newborns. Another purpose is to see what levels of SQV, low-dose RTV, ZDV, and 3TC are found in mothers and what levels of ZDV and 3TC are seen in newborns. Another purpose of this study is to see whether SQV passes from mother to newborn and if it passes at a level that is safe for the newborn.

Although ZDV has been able to reduce the rate of transmission of HIV from mother to child, it may be possible to reduce it further by using a combination of anti-HIV drugs. This study adds SQV (a protease inhibitor [PI]) with RTV (another PI) and 3TC (a reverse transcriptase inhibitor) to the mother's ZDV regimen.

DETAILED DESCRIPTION:
Although administration of ZDV to mother-infant pairs has dramatically reduced perinatal HIV infection, the goal is to reduce it further to less than 2%. In order to achieve this, combination strategies need to be developed for 2 purposes: 1) to reduce the perinatal transmission rate to goal levels; and 2) to provide other combination therapies for HIV-infected mothers whose virus has become resistant to ZDV, who have a very high viral load, or who have previously transmitted HIV while on ZDV. This study adds 3TC (another reverse transcriptase inhibitor) and SQV (a protease inhibitor [PI]) [AS PER AMENDMENT 08/15/00: with low-dose RTV (another PI)] to the mother's ZDV regimen.

During the antepartum period, mothers receive SQV with [AS PER AMENDMENT 08/15/00: low-dose RTV plus] ZDV and 3TC. At onset of active labor, mothers receive loading doses of each of the study drugs, then receive study drugs for 12 weeks postpartum on the same schedule as during the antenatal period. Within 12 hours of delivery, infants begin receiving 3TC and ZDV and continue until 6 weeks of age. Mothers are followed until 12 weeks postpartum and babies are followed until 6 months of age. [AS PER AMENDMENT 02/09/99: For maternal dosing, 1 Combivir tablet (containing 3TC and ZDV) may be administered in place of the individual agents 3TC and ZDV. Patients who prematurely discontinue study treatment should continue to be followed for the duration of the study.]

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are 14 to 32 weeks pregnant.
* Are at least 13 years old (need consent of parent or guardian if under 18).

Exclusion Criteria

Patients may not be eligible for this study if they:

* Cannot take ZDV, 3TC, or higher doses of RTV. Women who are able to tolerate low doses of RTV may be eligible.
* Are pregnant with more than 1 baby. (This study has been changed so that a patient pregnant with more than 1 baby is not eligible.)
* Have pregnancy complications or have medical problems that put pregnancy at risk.
* Have an active opportunistic (HIV-related) infection and/or serious bacterial infection at study entry.
* Have chronic diarrhea.
* Abuse alcohol or drugs.
* Do not have access to a participating clinic or are not willing to be followed at the same clinic for the duration of the study.
* Have received certain antiretroviral (anti-HIV) drugs or are taking certain medications. (This study has been changed to increase enrollment. The eligibility criterion in earlier versions was more restrictive, and has been changed to include women receiving SQV [with or without RTV], 3TC, and ZDV for longer than 3 weeks if their pre-entry viral load is 400 copies/ml or less OR if they have a significant reduction in viral load within 90 days of the pre-entry visit.)
* Plan to breast-feed.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24
Dates: Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Zorrilla, Study Chair; Arlene Bardeguez, Study Chair; Jane Pitt, Study Chair; Russell Van Dyke, Study Chair
Locations (15):
- United States (14):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Miami / Jackson Memorial Hosp, Miami, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ Hosp, New Orleans, Louisiana
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Columbia Presbyterian Med Ctr, New York, New York
  - Duke Univ Med Ctr, Durham, North Carolina
  - Med Univ of South Carolina, Charleston, South Carolina
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan, Puerto Rico

REFERENCES:
- [Background] Acosta EP, Zorrilla C, Van Dyke R, Bardeguez A, Smith E, Hughes M, Huang S, Pitt J, Watts H, Mofenson L; Pediatric AIDS Clinical Trials Group 386 Protocol Team. Pharmacokinetics of saquinavir-SGC in HIV-infected pregnant women. HIV Clin Trials. 2001 Nov-Dec;2(6):460-5. doi: 10.1310/PUY3-5JWL-FX2B-98VU. PMID 11742433